CLINICAL TRIAL: NCT03030014
Title: Effect of Dental Educational Program on Oral Hygiene Status Among Institutionalized Deaf Children. A Randomized Controlled Trial.
Brief Title: Effect of Dental Educational Program on Oral Hygiene Status Among Institutionalized Deaf Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sohil Souod Ali Shaalan, researcher at pedodontic department faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SShaalan
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- educational programm (Experimental): Oral health education will be done for children and their care givers about various diseases affecting the oral cavity, the effects of bad oral hygiene and tooth decay, importance of tooth brushing, and correct methods of tooth brushing.
  Three follow up examination is assessed after one week, three weeks and six weeks using questionnaire for evaluation of participant satisfaction about oral health and using OHIS index for evaluating the effect of the dental educational program on the oral health status of deaf children.
  Interventions: Behavioral: educational programm
- no educational programm (Placebo Comparator): without educational program Three follow up examination is assessed after one week, three weeks and six weeks using questionnaire for evaluation of participant satisfaction about oral health and using OHIS index for evaluating the effect of the dental educational program on the oral health status of deaf children.
  Interventions: Other: no educational program

INTERVENTIONS:
Behavioral: educational programm — Oral health education will be done for children and their care givers about various diseases affecting the oral cavity, the effects of bad oral hygiene and tooth decay, importance of tooth brushing, and correct methods of tooth brushing.Three follow up examination is assessed after one week, three weeks and six weeks using questionnaire for evaluation of participant satisfaction about oral health and using OHIS index for evaluating the effect of the dental educational program on the oral health status of deaf children.
  Arms: educational programm
Other: no educational program — without oral health education will be done for children and their care givers about various diseases affecting the oral cavity, the effects of bad oral hygiene and tooth decay, importance of tooth brushing, and correct methods of tooth brushing.Three follow up examination is assessed after one week, three weeks and six weeks using questionnaire for evaluation of participant satisfaction about oral health and using OHIS index for evaluating the effect of the dental educational program on the oral health status of deaf children.
  Arms: no educational programm

SUMMARY:
assess the effect of dental educational program on oral hygiene among institutionalized hearing impaired and mute children in Cairo, Egypt.

DETAILED DESCRIPTION:
* Evaluate participants satisfaction regarding the dental educational program(learning teeth brushing technique)
* Measure the oral hygiene index simplified to the participants at a different follow up periods for assessing the effect of the dental educational program on oral hygiene.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 6-12 years with mixed dentition.
* Institutionalized Deaf children in Cairo, Egypt.

Exclusion Criteria:

* Children above the age of 12 years and below the age of 6 years
* Patient un able to give informed consent
* Patient suffering from any other type of disability such as (mental retardation, physically and mentally handicapped, .etc.)
* Medically compromised patient
* Patient who were absent in the day of examination

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 6 weeks
  this outcome will be assessed via questionnaire

SECONDARY OUTCOMES:
oral hygiene index simplified | 6 weeks